CLINICAL TRIAL: NCT06849245
Title: Measuring Whether Promotion of a Digital Social Intervention by Primary Care Healthcare Professionals and Subsequent Engagement With Online Peer Support Improves Health and Well-being of Patients With Asthma and is Cost-effective: a Randomised Controlled Trial
Brief Title: Εffectiveness of a Digital Social Intervention in Primary Care
Acronym: ADHOC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); City, University of London (Other); University of Cambridge (Other); University of Edinburgh (Other); University of Nottingham (Other); University of Surrey (Other); St George's, University of London (Other); Asthma UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 349517
Record Dates: First submitted 2025-01-27; First posted 2025-02-27 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Asthma Intermittent, Uncontrolled

STUDY DESIGN:
Intervention Model Description: A general practice-based healthcare professional will carry out the study-related consultation (see 'Arms and Interventions' section below) and randomise participants to either the intervention or control group. Healthcare professionals will open a separate REDCap database to obtain the (automatically-generated) group assignment for the patient - either intervention or control - and will deliver the rest of the consultation accordingly.
Masking Description: Masking is not possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm in the ADHOC Trial (about 300 patients randomised to the intervention arm) (Experimental): A general practice-based healthcare professional will carry out the consultation and randomise participants to either the intervention or control group. Healthcare professionals will open a separate REDCap database to obtain the (automatically-generated) group assignment for the patient - either intervention or control - and will deliver the rest of the consultation accordingly. The intervention will consist of a one-off, face-to-face consultation with a practice-based clinician, followed by engagement with the Asthma + Lung UK online health community. The intervention will be delivered at the general practice with which each participant is registered.
  Interventions: Behavioral: A digital social intervention by primary care clinicians
- Control arm (about 300 patients randomised to the control arm) (No Intervention): Control group patients will receive usual care alone, without any reference to online health communities and online peer support.

INTERVENTIONS:
Behavioral: A digital social intervention by primary care clinicians — * Signposting to the online health community by explaining different sections of the website.
  * Introducing norms and values for passive (just reading) and active (writing posts) participation.
  * Motivation for engagement with the online health community, emphasising that it could be used ad hoc (e.g. when feeling unwell, or when they need information or emotional support).
  * Problem solving with respect to any difficulties/concerns.
  * Signing patients up to the online health community, by explaining terms and conditions.
  * Explaining the differences between posting publicly and privately (public posts are shared with third parties whereas private messages to other users are not shared).
  * Collection of baseline measures. Data will be entered into the study's online database.
  Patients will leave the consultation with a leaflet summarising all procedural matters in relation to signing up with the online health community and a reminder of their username and password.
  Arms: Intervention arm in the ADHOC Trial (about 300 patients randomised to the intervention arm)

SUMMARY:
The goal of this study is to deliver a definitive randomised controlled trial to measure the effectiveness and assess cost-effectiveness of a digital social intervention for patients with asthma, composed of promoting engagement with online peer support in a primary care consultation, followed by engagement with online peer support for 12 months. The main questions/objectives this study aims to answer/address are:

* Does promoting engagement with an online health community in primary care help people with troublesome asthma to experience fewer asthma symptoms?
* To assess cost-effectiveness of the intervention (including quality of life, well-being, use of healthcare services etc); stakeholder satisfaction (patients and healthcare professionals) with the intervention; fidelity of protocol delivery; context in which positive outcomes can be triggered.

DETAILED DESCRIPTION:
Patients with troublesome asthma, from 50-70 UK general practices, who might consider seeking advice online will be identified through a short online survey. The survey will include an asthma control test (ACT) questionnaire, a question about the network of support they have with their asthma, whether they are members of another existing online health community and whether they would be interested in taking part in a research study involving engagement in an asthma online health community (if randomised to the intervention arm).

Patients meeting the eligibility criteria will be asked to attend a one-to-one consultation with a healthcare professional at their general practice, who will randomise them using a randomisation tool and subsequently deliver the intervention encouraging them to engage with the asthma online health community or provide usual primary care, respectively. Participants of the intervention arm will be given a username and password for the Asthma + Lung UK online health community and shown how to login to the online health community. Participants will be asked to complete an online questionnaire at this consultation and again 12 months later. The consultation should take 30-45 minutes and completing the data-collection questionnaire 12 months later should take around 10 minutes.

During the 12-month period after the consultation, patients will be phoned by members of the research team every 3 months to collect data through an ACT questionnaire as well as volume of asthma exacerbations and associated healthcare utiilisation (primary and secondary care attendances) within last 3 months. Monthly text messages will also be sent to participants in the intervention arm who have consented, reminding them to engage with the online health community. The final follow-up questionnaire will include questions about how well their asthma is controlled, anxiety and depression, taking their asthma medication, and quality of life. Subject to participants' consent, the investigators will also endeavour to extract data from healthcare records about asthma exacerbations and use of primary and secondary care health services during the 12-month follow-up period (for both control and intervention arm participants). This data will be obtained from 'Discovery' for practices in North-East London. 'Discovery' is a clinical partnership project in East London, run by the Clinical Effectiveness Group at Queen Mary University of London and setting out to link primary and secondary care records, by creating a single database. The Clinical Effectiveness Group extracts data in an anonymised format. For practices in other parts of the UK, NHS Digital will be used to obtain data from healthcare records, and respective protocols and policies will be followed.

Data on intervention arm participants' use of the Asthma + Lung UK OHC during the study period will be collected and analysed, subject to consent, including the amount of engagement (number of days, hours/day etc.), community/ies joined, number of logins, number of likes, and time spent on pages, as well as the content of any public posts made by participants (private messages sent on the OHC will not be accessed or analysed).

At the end of the 12-month follow-up period, one-to-one interviews will be carried out with approximately 25 of the participating patients and approximately 15 of the HCPs involved in the study. Exact numbers will be determined by the point of data saturation being reached, with further interviewees being recruited if necessary. A convenience sample of participants will be invited (by email/text/phone) to take part in this one-off interview, which will last around one hour. Interviews will be carried out by a member of the research team and take place remotely via an appropriate online platform (Zoom or Microsoft Teams). During the interview, participants will be asked a series of questions (from a pre-determined list) exploring their views about their involvement in the study. Interviews will be audio recorded (after securing participants' consent - relevant field in the consent form) for subsequent analysis.

ELIGIBILITY:
Inclusion Criteria:

To participate in the study, participants will need to:

* Be adult asthma patients (aged 18 to 99) who have expressed their interest in digital social interventions in the recruitment survey.
* Report troublesome asthma (i.e. an ACT score of less than 20) in the recruitment survey).
* Be competent to consent for themselves, as determined by the healthcare professional delivering the consultation.

There are no specific criteria for selecting participants for the exit interviews (a convenience sample of patients and clinicians will be used and recruitment will continue until data saturation).

Exclusion Criteria:

* Patients who are already members of the Asthma + Lung UK online health community or other asthma online health communities/Facebook groups (i.e. general use of social media will not prevent participation).
* Palliative or end of life patients.
* Patients receiving institutional long-term care (receiving total care in residential homes or living in nursing homes).
* Patients considered unsuitable to take part in the study by their general practitioners/nurses.

There are no specific criteria for selecting participants for the exit interviews (a convenience sample of patients and clinicians will be used and recruitment will continue until data saturation).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Control of asthma | Baseline and very three months in a 12 month follow-up period
  Control of asthma will be self-reported by patients through an Asthma Control Test (ACT) questionnaire; minimum value: 5, maximum value: 25; higher scores indicate better asthma control.

SECONDARY OUTCOMES:
Anxiety | Baseline and at the end of a 12 month follow-up period
  Anxiety will be self-reported by patients through a GAD-7 (Generalised Anxiety Disorder 7-item instrument) questionnaire; minimum value: 0, maximum value: 21; higher scores indicate higher levels of anxiety.
Depression | Baseline and at the end of a 12 month follow-up period
  Depression will be self-reported by patients through a PHQ-8 (8-item Patient Health Questionnaire depression scale) questionnaire; minimum value: 0, maximum value: 24; higher scores indicate higher levels of depression.
Self-efficacy | Baseline and at the end of a 12 month follow-up period
  Self-efficacy will be self-reported by patients through the General Self-Efficacy Scale; minimum value: 10, maximum value: 40; higher scores indicate more self-efficacy.
Health-related quality of life | Baseline and very three months in a 12 month follow-up period
  Health-related quality of life will be self-reported by patients through an EQ-5D-5L (European Quality of Life 5 Dimensions 5 Level Version) questionnaire; minimum value: -0.59, maximum value: 1; higher scores indicate better quality of life.
Adherence to medications | Baseline and at the end of a 12 month follow-up period
  Adherence to medications will be self-reported by patients through a MARS-10 (10-item Medication Adherence Rating Scale) questionnaire; munimum value: 0, maximum value: 10; higher scores indicate better medication adherence.
Number of asthma exacerbations over last 3 months | Baseline and very three months in a 12 month follow-up period
  Asthma exacerbations will be self-reported by patients through bespoke questions
Primary and secondary care use over last 3 months | Baseline and very three months in a 12 month follow-up period
  Care use will be self-reported by patients through bespoke questions
Cost-effectiveness in relation to use of online health communities (likely a Markov model), including resource requirements, and costs for development, moderation, governance, and clinical oversight of online health communities | Calculations/estimations at various time-points during a 12 month follow-up period
  Within-trial and long-term cost-effectiveness analyses of online health communities' enhanced management versus current standard of asthma management in UK primary care. Costs of online health communities, healthcare and other resource use will be evaluated using nationally-representative unit costs of primary and secondary healthcare services. The within-trial cost-effectiveness will be assessed as incremental cost per quality-adjusted life year gained. The long-term cost-effectiveness of the OHCs will be evaluated using a long-term asthma model. Results will be presented as incremental cost effectiveness ratios.
Amount of online health community engagement (for intervention arm participants) | End of a 12 month follow-up period
  Amount of engagement with the online health community will be self-reported by patients through a bespoke question
Type (passive versus active) of online health community engagement (for intervention arm participants) | End of a 12 month follow-up period
  Type of engagement with the online health community will be self-reported by patients through a bespoke question
Amount of time spent on the online health community (for intervention arm participants) | End of a 12 month follow-up period
  Amount of time spent on the online health community will be provided to the research team by the manager of the Asthma + Lung UK online health community
Number of communities joined (for intervention arm participants) | End of a 12 month follow-up period
  Number of communities joined will be provided to the research team by the manager of the Asthma + Lung UK online health community
Number of logins to the online health community (for intervention arm participants) | End of a 12 month follow-up period
  Number of logins will be provided to the research team by the manager of the Asthma + Lung UK online health community
Number of likes on pages/posts within the online health community platform (for intervention arm participants) | End of a 12 month follow-up period
  Number of likes will be provided to the research team by the manager of the Asthma + Lung UK online health community
Time spent on pages within the online health community (for intervention arm participants) | End of a 12 month follow-up period
  Time spent on pages will be provided to the research team by the manager of the Asthma + Lung UK online health community
Public posts of the participants of the intervention arm within the online health community | End of a 12 month follow-up period
  Public posts will be provided to the research team by the manager of the Asthma + Lung UK online health community
Time of each public post in the online health community by the intervention arm participants | End of a 12 month follow-up period
  Time of posts will be provided to the research team by the manager of the Asthma + Lung UK online health community
Discussion thread of each public post in the online health community by the intervention arm participants | End of a 12 month follow-up period
  Discussion threads of each post will be provided to the research team by the manager of the Asthma + Lung UK online health community
User details in each discussion thread in the online health community in which one of the intervention arm participants was involved | End of a 12 month follow-up period
  User details in each discussion thread will be provided to the research team by the manager of the Asthma + Lung UK online health community
Experience of patients participating in the study | End of a 12 month follow-up period
  Experiences of patients will be obtained via qualitative interviews with patients
Experience of clinicians carrying out the study-related consultations | End of a 12 month follow-up period
  Experiences of clinicians will be obtained via qualitative interviews with clinicians

CONTACTS AND LOCATIONS:
Overall Officials: Anna De Simoni, PhD, Principal Investigator — Clinical Reader in Primary Care Research, Queen Mary University of London
Locations (5):
- United Kingdom (5):
  - South West Peninsula Regional Research Delivery Network, Exeter
  - East Midlands Regional Research Delivery Network, Leicester
  - North London Regional Research Delivery Network, London
  - North East and North Cumbria, Newcastle upon Tyne
  - East of England Regional Research Delivery Network, Norwich

IPD SHARING:
Plan to Share IPD: No
Data from individual participants will not be shared. Participants will not be individually identifiable from any research outputs. 'Pseudonymisation of data' will be the policy for ensuring confidentiality. All participants will be coded, by allocating them unique participation codes. The association between participation codes and names will be contained on a Word/Excel document and will be stored on a password-protected computer at Queen Mary University of London. Any electronic documents or hard copies of data collected from participants will only be accessible to the research team. Only members of the research team will have access to associations between names and participation codes. Every attempt will be made to pool/aggregate or coarsely categorise potentially identifiable information in any dissemination of research findings.

REFERENCES:
- [Background] Karampatakis GD, Wood HE, Griffiths CJ, Taylor SJC, Toffolutti V, Bird VJ, Lea NC, Ashcroft RE, Day B, Coulson NS, Panzarasa P, Li X, Sheikh A, Relton C, Sastry N, Watson JS, Marsh V, Mant J, Mihaylova B, Walker N, De Simoni A. Non-randomised feasibility study testing a primary care intervention to promote engagement in an online health community for adults with troublesome asthma: protocol. BMJ Open. 2023 Jul 11;13(7):e073503. doi: 10.1136/bmjopen-2023-073503. PMID 37433727
- [Background] Karampatakis GD, Wood HE, Griffiths CJ, Lea NC, Ashcroft RE, Day B, Walker N, Coulson NS, De Simoni A. Ethical and Information Governance Considerations for Promoting Digital Social Interventions in Primary Care. J Med Internet Res. 2023 Sep 27;25:e44886. doi: 10.2196/44886. PMID 37756051
- [Background] Karampatakis GD, Kimber S, Wood HE, Griffiths CJ, Taylor SJC, Li X, Day B, Mant J, Relton C, Watson JS, Marsh V, Coulson NS, De Simoni A. Development of the face-to-face component and recruitment strategy of a primary care digital social intervention for patients with asthma: Qualitative focus groups and interviews with stakeholders. Eur J Gen Pract. 2024 Dec;30(1):2407594. doi: 10.1080/13814788.2024.2407594. Epub 2024 Sep 27. PMID 39329323
- [Background] Karampatakis GD, Wood HE, Griffiths CJ, Taylor SJ, Toffolutti V, Bird VJ, Lea NC, Ashcroft R, Coulson NS, Panzarasa P, Li X, Sheikh A, Relton C, Sastry N, Watson JS, Mant J, Marsh V, Day B, Mihaylova B, Walker N, De Simoni A. Randomised controlled trial to measure effectiveness and cost-effectiveness of a digital social intervention promoted by primary care clinicians to adults with asthma to improve asthma control: protocol. BMJ Open. 2025 Sep 11;15(9):e104367. doi: 10.1136/bmjopen-2025-104367. PMID 40940055